CLINICAL TRIAL: NCT00529386
Title: A Prospective Pilot Study to Evaluate the Safety and Efficacy of Botox™ for the Treatment of Men Diagnosed With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Brief Title: Botox for Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Dr. J. Curtis Nickel, Principal Investigator, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOTOX-CP
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Prostatitis; Chronic Pain Syndrome
Keywords: prostatitis; Botox
MeSH Terms: conditions — Prostatitis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botox (Experimental): 300 IU botox
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — 300 units
  Other Names: Botulinem toxin

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of intraprostatic injection of Botox for the treatment of men diagnosed with chronic nonbacterial prostatitis/chronic pelvic pain syndrome (CP/CPPS).

DETAILED DESCRIPTION:
This is a prospective open label study examining the efficacy and safety of intraprostatic Botox . Men with a clinical diagnosis of chronic nonbacterial prostatitis/CPPS will be treated with intraprostatic Botox™ and followed for 12 weeks (primary efficacy analyses), and 24 weeks (long term follow-up) for responders.

It is proposed that a total of 40 males will be enrolled. There will be seven (7) research clinic visits and two phone contacts: Visit 1 (screening), Visit 2 (baseline/treatment), Visit 3 (2-week safety evaluation - clinic contact), Visit 4 (4-week safety evaluation - phone contact), Visit 5 (6-week interim efficacy/safety), Visit 6 (12-week primary endpoint evaluation), Visit 7 (14-week clinic follow up), Visit 8 (16 week phone contact) and Visit 9 (24-week clinic close out).

Outcome measures include Chronic Prostatitis Symptom Index (CPSI 0-35), NRS pain (0-10), Global Response Assessment (GRA) at 12 weeks. Safety to be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has signed and dated the appropriate Informed Consent document.
2. Participant must be ≥ 18 years of age.
3. Participant has had a clinical diagnosis of chronic nonbacterial prostatitis (chronic pelvic pain syndrome) (CPPS) defined as symptoms of discomfort or pain in the perineal or pelvic region for at least the past 3 months without evidence of bacterial infection.
4. Participants must report ejaculatory pain and/or perineal discomfort.
5. Participants must have pain or discomfort localized to perineum or prostate during physical examination.
6. Participants must have an aggregate score of greater than or equal to 15 on the National Institutes of Health chronic prostatitis symptom index (NIH-CPSI).
7. Participant must have > 8 on the pain domain sub-score of the NIH-CPSI.
8. Participant must have had empiric treatment with 4 weeks fluoroquinolone, and subsequently failed the antibiotic therapy.

Exclusion Criteria:

1. Participant has a history of prostate, bladder or urethral cancer.
2. Participant has inflammatory bowel disease (such as Crohn's disease or ulcerative colitis, but not irritable bowel syndrome).
3. Participant has undergone pelvic radiation or systemic chemotherapy.
4. Participant has undergone intravesical chemotherapy.
5. Participant has been treated for unilateral orchialgia without pelvic symptoms.
6. Participant has a current urethral stricture and/or bladder stones.
7. Participant has a neurological disease or disorder affecting the bladder.
8. Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.
9. Participant has a documented UTI within the last 3 months.
10. Participant has evidence of facultative Gram negative or enterococcus with a value of ≥ 1000 CFU/ml in mid-stream urine (VB2).
11. Participant has had previous intraprostatic injection of Botox.
12. Participant currently enrolled in an investigational study.
13. Participant interested in future fertility/fathering children.
14. Participant with urinary retention (PVR >200cc).
15. Participant having had prostate surgery in the past 3 months.
16. Participant having had minimally invasive surgical therapy for BPH.
17. Participant with a cystostomy or nephrostomy.
18. Participant with penile or urinary sphincter implants.
19. Participant with previous rectal surgery, current rectal disease or peri-rectal inflammatory disorders except hemorrhoidectomy.
20. Participant with PSA >10 ng/ml(PSA range 4-10, biopsy at PI discretion (deferral).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Curtis Nickel, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Advanced Urological Research, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botox
Started | 7 (Study has been discontinued)
Completed | 6 (Study discontinued after 7 patients enrolled and analyzed)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Botox
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants] — CPSI range for CP/CPPS
  Participants
    <=18 years | 0
    Between 18 and 65 years | 7
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: GRA
Description: At 12 weeks there were no GRA responders. Study stopped because of futility.
Time Frame: 12 weeks
Population: 7 CPCPPS patients enrolled and analysed before stopping study because of futility
Measure: Count of Participants; unit: Participants
Arm/Group | Botox
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Arm/Group | Botox
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No